CLINICAL TRIAL: NCT05534087
Title: A Randomized Controlled Phase III Trial of Treatment Intensification in Stage II-III Colon Cancer Patients With Positive MRD During Adjuvant Chemotherapy
Brief Title: Platform Study of Circulating Tumor DNA Directed Adjuvant Chemotherapy in Colon Cancer (KCSG CO22-12)
Acronym: CLAUDIA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sae-Won Han, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2205-029-1322
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Colon Cancer
Keywords: Minimal residual disease; Intensified chemotherapy
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm, Residual | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mFOLFIRINOX intensified chemotherapy (Experimental): 6 cycles of mFOLFIRINOX
  - Modified FOLFIRINOX (mFOLFIRINOX) regimen: 6 cycles every 2 weeks
  Interventions: Drug: mFOLFIRINOX-FOLFIRI intensified chemotherapy
- FOLFOX or CAPOX adjuvant chemotherapy (Active Comparator): FOLFOX 6 cycles or CAPOX 4 cycles
  * FOLFOX regimen: 6 cycles every 2 weeks or
  * CAPOX regimen: 4 cycles every 3 weeks
  Interventions: Drug: FOLFOX or CAPOX adjuvant chemotherapy

INTERVENTIONS:
Drug: mFOLFIRINOX-FOLFIRI intensified chemotherapy — (1) Modified FOLFIRINOX (mFOLFIRINOX) regimen: 6 cycles every 2 weeks
  * Oxaliplatin 85mg/m2 IV infusion over 120 min D1
  * Leucovorin 400mg/m2 IV (concurrently with oxaliplatin)
  * Irinotecan 150mg/m2 IV infusion over 60-90 min D1
  * 5-fluorouracil 2,400mg/m2 IV infusion continuously over 46-48h D1-2
  Arms: mFOLFIRINOX intensified chemotherapy
Drug: FOLFOX or CAPOX adjuvant chemotherapy — 1. FOLFOX regimen: 6 cycles every 2 weeks
     * Oxaliplatin 85mg/m2 IV infusion over 120 min D1
     * Leucovorin 400mg/m2 IV infusion over 120 min (concurrently with oxaliplatin)
     * 5-fluorouracil 400mg/m2 IV bolus D1
     * 5-fluorouracil 2,400mg/m2 IV infusion continuously over 46-48h D1-2 or
  2. CAPOX regimen: 4 cycles every 3 weeks
     * Oxaliplatin 130mg/m2 IV infusion over 120 min D1
     * Capecitabine 1,000mg/m2 PO bid D1-14
  Arms: FOLFOX or CAPOX adjuvant chemotherapy

SUMMARY:
This study is a prospective, open-label, randomized phase 3 clinical trial. It aims to investigate if the early introduction of intensified chemotherapy (3 months of modified FOLFIRINOX) improves the 3-year disease-free survival rate compared to standard treatment (FOLFOX/CAPOX for an additional three months to complete six months of standard adjuvant chemotherapy) in patients with stage 2-3 colon cancer in whom ctDNA MRD in the part 1 study remained positive during adjuvant FOLFOX/CAPOX chemotherapy

DETAILED DESCRIPTION:
About 25% of resectable high-risk stage 2 or stage 3 colon cancers are known to relapse despite standard treatments, including radical resection and adjuvant chemotherapy.

Using circulating tumor DNA (ctDNA)-based minimal residual cancer (MRD) detection technology, patients whose MRD is not eradicated after adjuvant chemotherapy could be identified. Early introduction of intensified chemotherapy for this group of patients could prolong survival time and increase cure rates.

This study is part of the Platform Study of Circulating Tumor DNA Directed Adjuvant Chemotherapy in Colon Cancer (CLADIA Colon Cancer). Part 1 of the platform study (Prospective Observational Study of ctDNA Monitoring During Adjuvant) is a large-scale, prospective observational study that follows ctDNA up to three years after resection in about 1,200 patients with stage 2-3 colon cancer.

This study (Part 2) aims to study the efficacy of early intensified chemotherapy (3 months of modified FOLFIRINOX ) compared to standard treatment (FOLFOX/CAPOX for an additional three months to complete six months of standard adjuvant chemotherapy) in patients with stage 2-3 colon cancer in whom ctDNA MRD in the part 1 study remained positive during adjuvant FOLFOX/CAPOX chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who willingly consented and signed the informed consent form to participate in the study
2. Age range of 19 to 75 years
3. Adenocarcinoma of colon confirmed by histology
4. Patients with stage II-III colon cancer as defined by the American Joint Committee on Cancer's eighth edition (Stage II cancer is limited to patients who are at a high risk, with more than one risk factor for recurrence.)
5. Patients who have completed the sixth cycle of FOLFOX or the fourth cycle of CAPOX adjuvant chemotherapy for colon cancer following radical resection (R0 resection)
6. A ctDNA test performed 3 to 6 weeks after surgery reveals a positive MRD
7. ECOG performance scale of 0-1 (only 1 is allowed for 70-75 years old)
8. Adequate bone marrow function [ANC ≥1,300/LL, platelets ≥75,000/LL, hemoglobin ≥8.0g/dL (may be eligible in study if intermittent transfusion is required)]
9. Appropriate liver function (total bilirubin ≤1.5xULN, AST and ALT ≤3xULN)
10. Appropriate renal function (serum creatine ≤1.5xULN, renal clearance rate ≥50 ml/min)
11. Patients who are deemed to understand the study protocol and are willing to participate in the trial until it is completed

Exclusion Criteria:

1. Pregnant or lactating women
2. Pregnant women who had a positive pregnancy test at the time of the baseline examination (postmenopausal women must be amenable for at least 12 months to be considered non-fertility)
3. Sexually active men and women of reproductive age who are unwilling to use contraception throughout the study treatment and for a period of 6 months (female) or 3 months (male) following the discontinuation of study treatment
4. Clinically significant heart condition [unstable angina requiring medication, symptomatic coronary artery disease, congestive heart failure, or significant heart arrhythmia above NYHA II, or acute coronary syndrome, including myocardial infarction within the last 6 months]
5. Active viral infections such as HIV (However, HBV carriers may enroll if their HBV DNA titer is less than 20,000 IU/ml, and antiviral drugs for hepatitis B may be administered prophylactically at the investigator's discretion)
6. Significant uncontrolled infections or other uncontrolled comorbidities
7. Symptomatic inflammatory bowel disease
8. Allogeneic transplantation history necessitating immunosuppressive therapy
9. A history of other malignancies identified within the last three years, except for completed removed basal cell carcinoma of the skin, completely removed cervical epithelial carcinoma, and thyroid cancer that has been treated, including surgery
10. Recurrent or residual disease identified clinically or radiographically
11. Previous history of irinotecan treatment
12. Polyposis including familial adenomatous polyps
13. Two or more colon or rectal cancers with a pathologic stage greater than II that were detected concurrently or within the last three years
14. When the investigator determines that the subjects' safety may be jeopardized during the study because of other serious or unstable pre-existing medical or mental conditions
15. Prior clinical trial participation and usage of investigational drugs or devices following radical resection of colon cancer
16. Patients with peripheral neuropathy who have a CTCAE v5 grade 3 or higher functional disability (corresponds to "severe symptoms, limiting self-care activity of daily living" according to CTCAE v5 criteria)
17. Previous anaphylactic reaction or severe and unexpected reactions to fluoropyrimidines or platinum
18. Gilbert's syndrome, dehydro-pyridine dehydrogenase (DPD) deficiency, or homozygous UGT1A1*28 alleles

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival rate | Through completion of follow-up (estimated to be 36 months)
  The rate refers to cases that see first tumor metastasis or recurrence or death of any cause from randomization

SECONDARY OUTCOMES:
Circulating tumor DNA (ctDNA) clearance rate | The data of ctDNA clearance rate will be collected at 10 time points
  The proportion of patients with circulating tumor DNA clearance after 36months study treatment.
5-year overall survival rate (5y-OS rate) | Through completion of follow-up (estimated to be 60 months)
  Overall survival is defined as the time from beginning of study treatment until death due to any cause.
Treatment-Related Adverse Events | Through completion of follow-up (estimated to be 36 months)
  The number of patients with adverse events and the severity according to CTCAE v5.0.
EORTC QLQ-C30 scale | Through completion of follow-up (estimated to be 36 months)
  Using the EORTC QLQ-C30 scale (European Organization for Research on Treatment of Cancer Quality of Life Questionnaire-Core 30) to evaluate the quality of life of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sae-Won Han, MD,PhD, Principal Investigator — Seoul National University Hospital South Korea; Youngjun Cha, MD, Study Director — Natioal Cancer Center South Korea
Locations (3):
- South Korea (3):
  - National Cancer Center, Goyang
  - Jin Won Kim, Seongnam
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No